CLINICAL TRIAL: NCT06960954
Title: Prothrombin Induced by Vitamin K Absence II (PIVKA-II) Serum Level as a Predictor for Portal Vein Tumor Thrombosis in Hepatocellular Carcinoma Patients.
Brief Title: PIVKA-II for Predicting Portal Vein Thrombosis in Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical medicine, Tanta University
Other Study IDs: 36264PR1127/3/25
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hepato Cellular Carcinoma (HCC); Portal Vein Tumour Thrombosis
Keywords: PIVKA-II; Portal vein tumor thrombosis; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC patients with PVTT.: 58 HCC patients with PVTT.
  Interventions: Diagnostic Test: Prothrombin induced by vitamin K absence II (PIVKA-II)
- HCC Patients without PVTT.: 58 HCC Patients without PVTT.
  Interventions: Diagnostic Test: Prothrombin induced by vitamin K absence II (PIVKA-II)

INTERVENTIONS:
Diagnostic Test: Prothrombin induced by vitamin K absence II (PIVKA-II) — Serum PIVKA-II level will be measured in HCC patients with and without PVTT.

SUMMARY:
The goal of this cross-sectional observational study is to evaluate the relation between Prothrombin induced by vitamin K absence II (PIVKA-II) and the presence of portal vein tumor thrombosis (PVTT) in hepatocellular carcinoma (HCC) patients.

Researchers will compare PIVKA-II serum levels in HCC patients with PVTT and without PVTT.

Participants will undergo history-taking, clinical examination, laboratory investigations, PIVKA-II serum level, Child-Pugh classification, Model for End-stage Liver Disease (MELD) score, BCLC staging, abdominal ultrasonography, and Triphasic CT abdomen with contrast or MRI to evaluate tumor site, size, number, and presence of PVTT (a filling defect in the portal vein or its branch to distinguish PVTT or thrombus).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years.
* Patients with confirmed HCC with or without PVTT (Diagnosed by two imaging modalities or one imaging modality with elevated serum alpha fetoprotein or liver biopsy).

Exclusion Criteria:

* Prior locoregional therapy or liver transplantation.
* Patients on vitamin K, vitamin K antagonists or antibiotics.
* Patients with cholestasis.
* Patients with renal insufficiency.
* Patients with other malignancies.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will be carried out on 116 patients attending the Tanta Tropical Medicine Outpatient Clinic, Faculty of Medicine. The start of the research will be in January 2025 to December 2025 or until the collection of the cases.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PIVKA-II serum level for prediction of PVTT in HCC patients. | through study completion, an average of 1 year
  PIVKA-II level (mAU/mL) will be measured in serum of HCC patients with and without PVTT.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Elkafoury, MD, Study Director — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt